CLINICAL TRIAL: NCT01753232
Title: Non-interventional Study: Safety and Efficacy of the DALI LDL-adsorber and MONET-lipoprotein Filter
Brief Title: Safety and Efficacy of the DALI LDL-adsorber and MONET Lipoprotein Filter
Acronym: LINET
Status: Completed | Type: Observational
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: TA-DALI-MONET-01-D
Record Dates: First submitted 2012-12-13; First posted 2012-12-20 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Hypercholesterolemia, Familial; LIPOPROTEIN TYPES--Lp SYSTEM Lp(a) HYPERLIPOPROTEINEMIA
Keywords: DALI adsorber; MONET lipoprotein filter
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Lipoprotein Types--Lp System Lp(A) Hyperlipoproteinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DALI-adsorber, hypercholesterolemia: Patients suffering from familial hypercholesterolemia treated at least twice a month with the DALI-system
  Interventions: Device: DALI-adsorber
- MONET-Filter, hypercholesterolemia: Patients suffering from familial hypercholesterolemia treated with the MONET-Lipoprotein filter
  Interventions: Device: MONET-Lipoprotein filter

INTERVENTIONS:
Device: DALI-adsorber — Recording of treatment data. No extra interventional treatment
  Groups: DALI-adsorber, hypercholesterolemia
Device: MONET-Lipoprotein filter — Only treatment data recording. No extra interventional treatment
  Groups: MONET-Filter, hypercholesterolemia

SUMMARY:
Low Density Lipoprotein (LDL)-apheresis refers to a procedure in which blood taken from a patient's vein is cleaned from pathogenic substances, e.g. cholesterol, outside the body and then given back to the patient. In the DALI (Direct Adsorption of Lipoproteins)-system whole blood is pumped over an adsorber containing beads that selectively bind LDL-cholesterol. The MONET (Membrane filtration Optimized Novel Extracorporeal Treatment)-system works with plasma which is cleaned by filtration. This study comprises the recording of safety and efficacy data from patients treated either with the DALI or MONET-system over a period of 2 years.

DETAILED DESCRIPTION:
Data were recorded from patients suffering from familial hypercholesterolemia and treated by lipid apheresis using one of the two systems investigated for at least 3 months prior to inclusion in the study. Only those treatments were documented in which routine blood samples for laboratory analysis were taken, or in which adverse or serious adverse device effects occur.

ELIGIBILITY:
Inclusion Criteria:

* given informed consent
* 18 years or older
* patient compliant to therapy as prescribed
* at least two therapy sessions per month
* treatment with DALI or MONET system for at least 3 months before inclusion
* last severe invasive intervention in hospital more than 3 months ago

Exclusion Criteria:

* earlier participation in the study
* unconscious patient/persons without capacity to contract
* for DALI: intake of ACE-inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypercholesterolemic patients from free-standing private apheresis centres and one hospital department
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change of Low Density Lipoprotein (LDL)-Concentration | Every two weeks to every three months for 24 months
  Data are only recorded for visits with lab results

SECONDARY OUTCOMES:
Blood/plasma volume treated | Every two weeks to every three months for 24 months
Number of occurence of adverse and serious adverse device effects | 24 months
Change of Lipoprotein(a)-concentration | Pre/post treatment over 24 months, once per month or every 3 months
  Only in patients with isolated Lp(a) increase
Change of total cholesterol | Every two weeks to every three months for 24 months
  Only for treatment sessions with lab results
Change of High Density Lipoprotein (HDL)-concentration | Every two weeks to every three months for 24 months
  Only for treatment sessions with lab results
Change of triglyceride-concentration | Every two weeks to every three months for 24 months
  Only for treatment sessions with lab results
Change in blood count | Every two weeks to every three months for 24 months
  Only for treatment sessions with lab results
Change of fibrinogen-concentration | Every two weeks to every three months for 24 months
  Only for treatment sessions with lab results
Change of creatinine-concentration | Every two weeks to every three months for 24 months
Change of Immunoglobulins (Ig) | Every two weeks to every three months for 24 months
  Only for treatment sessions with lab results, Immunoglobulin (Ig) G, IgA and IgM if measured. In MONET patients only.
Change in C Reactive Protein (CRP)-concentration | Every two weeks to every three months for 24 months
  Only for treatment sessions with lab results
Change of blood pressure and heart rate | Every two weeks to every three months for 24 months
  Only for treatment sessions with lab results
Blood or plasma flow | Every two weeks to every three months for 24 months
Anticoagulation regime | Every two weeks to every three months for 24 months
Treatment time | Every two weeks to every three months for 24 months
Medication | Every two weeks to every three months for 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Heinzler, MD, Principal Investigator — Gemeinschaftspraxis Gysan, Heinzler, May, Hossmann; Franz Heigl, MD, Principal Investigator — Dres. Heigl, Hettich & Partner Medizinisches Versorgungszentrum; Frank Leistikow, MD, Principal Investigator — Nierenzentrum Mannheim; Frido Himmelsbach, MD, Principal Investigator — Apheresezentrum Ingelheim; Ralf Spitthöver, MD, Principal Investigator — Nephrologische Gemeinschaftspraxis Dialysezentrum/Lipidzentrum; Eberhard Roeseler, MD, Prof, Principal Investigator — Zentrum für Nieren,- Hochdruck und Stoffwechselerkrankungen Standort Heidering; Volker Schettler, MD, Principal Investigator — Nephrologisches Zentrum Goettingen; Gerd Schmitz, MD, Prof, Principal Investigator — University Regensburg Department Clinical Chemistry and Laboratory Medicine; Nadim Abduhl-Rahman, MD, Principal Investigator — Dialysezentrum Magdeburg-Stadtfeld; Jens Ringel, MD, Principal Investigator — Dialysezentrum Potsdam; Wolfgang Ramlow, MD, Principal Investigator — Apheresezentrum Rostock
Locations (11):
- Germany (11):
  - Nierenzentrum Mannheim, Mannheim, Baden Würtemberg
  - Medizinisches Versorgungszentrum, Kempten (Allgäu), Bavaria
  - Universitätsklinikum Regensburg Institut für Klinische Chemie und Laboratoriumsmedizin, Regensburg, Bavaria
  - Dialysezentrum Potsdam, Potsdam, Brandenburg
  - Nephrologisches Zentrum Goettingen, Göttingen, Lower Saxony
  - Zentrum für Nieren und Hochdruckkrankheiten Standort Heidering, Hanover, Lower Saxony
  - Apheresezentrum Rostock, Rostock, Mecklenburg-Vorpommern
  - Gemeinschaftspraxis Gysan, Heinzler, May, Hossmann, Cologne, North Rhine-Westphalia
  - Nephrologische Gemeinschaftspraxis Dialysezentrum/Lipidzentrum, Essen, North Rhine-Westphalia
  - Apheresezentrum Ingelheim, Ingelheim, Rhineland-Palatinate
  - Dialysezentrum Magdeburg-Stattfeld, Magdeburg, Saxony-Anhalt